CLINICAL TRIAL: NCT02511808
Title: Adaptive Interventions for Problem Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Jonathan Morgenstern, Director, Addiction Services, Northwell Health
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 14-413; R01AA022714 (NIH)
Record Dates: First submitted 2015-07-10; First posted 2015-07-30 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Alcohol-Related Disorders; Alcohol Use Disorders; Alcohol Drinking; Alcoholism; Alcohol Abuse
Keywords: Drinking; Alcohol Problems; Alcoholism; Reduced Drinking; Problematic Drinking; Non-Abstinence-based Drinking; Controlled Drinking; Heavy Drinking
MeSH Terms: conditions — Alcohol-Related Disorders; Alcoholism; Alcohol Drinking | interventions — Crisis Intervention; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Step-up Treatment: MI (Active Comparator): After receiving one session of Brief Advice (BA), participants will be assessed at week 4 for response to this treatment. Those who are deemed non-responders to the BA will be randomly assigned to receive either Motivational Interviewing (MI) or more BA. In this arm, participants will receive two sessions of MI.
  Interventions: Behavioral: Motivational Interviewing
- Control: BA (Other): After receiving one session of Brief Advice (BA), participants will be assessed at week 4 for response to this treatment. Those who are deemed non-responders to the BA will be randomly assigned to receive either Motivational Interviewing (MI) or more BA. In this arm, participants will receive one additional session of BA.
  Interventions: Behavioral: Brief Advice
- Step-up Treatment: Specialist Care (Active Comparator): After receiving one session of Brief Advice (BA) and two sessions of Motivational Interviewing (MI) or one session of BA over the first 8 weeks of the study, participants will be assessed at week 8 for response to this treatment. Those who are deemed non-responders will be randomly assigned to receive Behavioral Self-Control Training (BSCT) or more MI if they were randomized to MI at week 4 or five sessions of combined MI and BSCT or one more session of MI if they were randomized to BA at week 4. In this arm, participants will receive four sessions of BSCT if they received MI at the previous randomization or five sessions of combined MI and BSCT if they received BA at the previous randomization.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Behavioral Self-Control Training
- Control: MI (Other): After receiving one session of Brief Advice (BA) and two sessions of Motivational Interviewing (MI) or one session of BA over the first 8 weeks of the study, participants will be assessed at week 8 for response to this treatment. Those who are deemed non-responders will be randomly assigned to receive Behavioral Self-Control Training (BSCT) or more MI if they were randomized to MI at week 4 or five sessions of combined MI and BSCT or one more session of MI if they were randomized to BA at week 4. In this arm, participants will receive one session of MI if they received MI at the previous randomization or two sessions of MI if they received BA at the previous randomization.
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Brief Advice — Brief Advice (BA) consists of a 20-minute session delivered by a study therapist, adhering to the NIAAA's Clinician Guide to Problem Drinkers. It includes personalized, normative feedback based on NIAAA drinking norms, goal selection, instructions on self-monitoring, discussion of drink reduction strategies, and distribution of the NIAAA bibliotherapy guide.
  Arms: Control: BA
Behavioral: Motivational Interviewing — Motivational Interviewing will consist of standard techniques, such as developing discrepancy, enhancing motivation, and developing a change plan, that have been adapted to treatment for problem drinkers.
  Arms: Control: MI; Step-up Treatment: MI; Step-up Treatment: Specialist Care
Behavioral: Behavioral Self-Control Training — Behavioral Self-Control Training will consist of Cognitive Behavioral Therapy adapted to problem drinkers, whose core components include a functional analysis, skills training, daily self-monitoring, homework, and graded exposures and mastery of high risk situations.
  Arms: Step-up Treatment: Specialist Care

SUMMARY:
The purpose of this study is to understand how certain interventions help people reduce or quit their drinking and how certain interventions may help best at certain points in time in the change process.

DETAILED DESCRIPTION:
Problem drinkers (PDs) represent a majority of the estimated 32 million Americans with alcohol problems that spans a spectrum of severity from individuals who drink excessively and experience of occasional negative consequences to those with moderate Alcohol Dependence (AD) and intact psychosocial functioning. PDs can benefit from relatively brief treatment that could be delivered in mainstream healthcare, but less than 5% receive such care. In addition, PD treatment is only modestly effective, and there is a surprising absence of empirical research to guide PD treatment selection. Adaptive Interventions (AI) are a novel approach to treatment development that may have significant advantages over fixed treatments in improving efficacy and fostering adoption of Evidence Based Practices in mainstream healthcare. If study aims are achieved, a set of empirically-derived decision support tools will be created to guide Alcohol Use Disorders (AUD) care similar to tools that exist for other chronic diseases. In addition, new knowledge will be gained about Mechanisms of Behavior Change of AUD that can guide future AUD treatment research. Finally, important progress will be made in methods that capitalize on the remarkable advances in sensor technologies, advanced mathematics, and engineering to create a new type of tailored, near-real time feedback, adaptive behavior therapies.

ELIGIBILITY:
Primary Inclusion Criteria: Adults who have heavy weekly alcohol consumption (and/or an alcohol use disorder) and are willing to reduce their drinking.

Primary Exclusion Criteria: Adults for whom the level of treatment provided is not appropriate and/or who require more intensive substance use or psychiatric treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Time Line Follow Back | 24 Weeks
  Calendar-based method of recording drinking patterns. Data will be aggregated into summary variables.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Morgenstern, Ph.D., Principal Investigator — Northwell Health; Nehal P Vadhan, Study Director — Northwell Health
Locations (1):
- Northwell Health, Great Neck, New York, United States

REFERENCES:
- [Background] Kuerbis AN, Shao S, Treloar Padovano H, Jadanova A, Selva Kumar D, Vitale R, Nitzburg G, Vadhan NP, Morgenstern J. Context and craving among individuals with alcohol use disorder attempting to moderate their drinking. Exp Clin Psychopharmacol. 2020 Dec;28(6):677-687. doi: 10.1037/pha0000349. Epub 2020 Jan 23. PMID 31971419